CLINICAL TRIAL: NCT00687362
Title: A Multicenter, Multinational, Open Label Study on the Efficacy and Safety of Infliximab Monotherapy in Moderate-to-severe Chronic Plaque Psoriasis in Middle Eastern Population
Brief Title: A Study to Evaluate Remicade (Infliximab) in Moderate-to-Severe Chronic Plaque Psoriasis in the Middle Eastern Population (Study P04528)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04528
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infliximab 5 mg/kg (Experimental): Infliximab 5 mg/kg of body weight given as an infusion at Weeks 0, 2, 6, 14, and 22.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab 5 mg/kg of body weight given as an infusion at Weeks 0, 2, 6, 14, and 22.
  Other Names: Remicade, SCH 215596

SUMMARY:
Middle Eastern subjects with moderate-to-severe chronic plaque psoriasis will be administered infusions of infliximab (Remicade) at 5 mg/kg of body weight at Weeks 0, 2, 6, 14, and 22. The safety and efficacy of infliximab monotherapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, either gender, and any race.
* Psoriasis affecting >=5% of body surface, PASI score >=10 (maximum score 72).
* History of plaque psoriasis for >6 months.
* Informed written consent.
* Refractory to other anti-psoriasis agents (topical corticosteroids, phototherapy UVa [PUVA], or systemic therapy).
* Negative chest x-ray and purified protein derivative (PPD) within 1 month.
* Understand and be able to adhere to dosing and visit schedules.
* Screening laboratory tests must meet protocol-specified criteria.
* Women and men of childbearing potential must be using adequate birth control measures and should continue such precautions for 6 months after last infusion of infliximab.

Exclusion Criteria:

* Pregnant, nursing, or planned pregnancy within 6 months after last scheduled treatment.
* Used topical corticosteroids in previous 14 days or systemic therapy (phototherapy UVb [UVB], PUVA, cyclosporine, methotrexate) in previous 28 days, or received treatment with anti-tumor necrosis factor (TNF)-alpha monoclonal antibodies, human or murine immunoglobulins, TNF-alpha receptor fusion proteins, or other bioengineered fusion proteins.
* Received previous immunobiologics.
* Have HIV, hepatitis B or C.
* Recently transplanted (exception - corneal transplant >3 months prior to first infusion) or known malignancy or history of malignancy within previous 5 years (exception - basal or squamous cell carcinoma of skin that has been treated with no evidence of recurrence).
* Concurrent medications that are not permitted.
* congestive heart failure (CHF)
* Use of cyclosporine or tacrolimus within 4 weeks prior to Screening.
* Use of intramuscular (IM), intravenous (IV), or oral corticosteroids within 4 weeks prior to Screening.
* Treatment with any investigational drug within 3 months prior to Screening.
* Allergy to murine proteins.
* Serious infections (hepatitis, pneumonia, pyelonephritis) in previous 3 months.
* History of active tuberculosis (TB) requiring treatment within previous 3 years, or history of opportunistic infections (herpes zoster) within 2 months of Screening.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurological or cerebral disease.
* Current signs or symptoms of other severe uncontrolled disease which in investigator's opinion would put the subject at an unacceptable risk.
* History of current alcohol or drug abuse.
* Not observed designated washout periods for any of the prohibited medications in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-05-30 (Actual); Primary Completion 2008-11-11 (Actual); Study Completion 2008-11-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infliximab 5 mg/kg
Started | 22
Completed | 19 (Completed protocol at Week 24)
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.05 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 19
Region of Enrollment [Number; unit: participants]
  Middle East | 22

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index 75 (PASI75) Response at Week 10
Description: PASI 75 response is defined as participants who achieved at least a 75% improvement in PASI score from Baseline to Week 10.
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 to 72 (the higher the number, the worse the disease).
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 22
participants | 16

ADVERSE EVENTS:
Arm/Group | Infliximab 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 11/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg (N=22)
vomiting (Gastrointestinal disorders) | 3 (3)
pyrexia (General disorders) | 4 (5)
tinea versicolour (Infections and infestations) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
psoriasis (Skin and subcutaneous tissue disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees not to publish/publicly present any interim results of the Study without prior written consent of Sponsor. The PI further agrees to

provide 30 days written notice to Sponsor prior to submission for publication/presentation to allow Sponsor to review materials which report any results of the Study. Sponsor shall have the right to review/comment on

any presentation, which include editorial rights to ensure protection of confidential information, accuracy, and fair balance.